CLINICAL TRIAL: NCT03074370
Title: Evaluation of Smile Esthetics in Orthodontically Treated Adult Female Patients With Bimaxillary-dentoalveolar Protrusion: A Retrospective Cohort Study
Brief Title: Evaluation of Smile Esthetics in Orthodontically Treated Patients With Bimaxillary-dentoalveolar Protrusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Abo elnaga, Principal Investigator, Cairo University
Other Study IDs: CEBC-CU-2017-02-08
Record Dates: First submitted 2017-02-25; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Bimaxillary Protrusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of Smile Esthetics in Orthodontically Treated Adult Female Patients with Bimaxillary-dentoalveolar Protrusion.

A Retrospective Cohort Study.

ELIGIBILITY:
The selected records should meet the following inclusion criteria:

Pre treatment:

1. Full permanent dentition
2. No dental nor any craniofacial anomalies
3. Molar Class I with bimaxillary-dentoalveolar protrusion
4. No excessive over jet or overbite

Treatment mechanics:

1. All patients treated with extraction of four 1st premolars
2. Retraction of anterior teeth using maximum anchorage mechanics

Post treatment:

1. Canine 1 relation
2. Molar I relation

Exclusion criteria :

Any orthodontic records without the previously mentioned pre and posttreatment inclusion criteria

Ages: 14 Years to 24 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Adult Egyptian females with bimaxillary-dentoalveolar protrusion.
Study Population: Study models of orthodontically treated Egyptian adult female patients with bimaxillary dentoalveolar protrusion .
Sampling Method: Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Gingival display | Change from Baseline gingival display, at an average 24 months
  Amount of maxillary gingival exposure between inferior border of upper lip and marginal gingiva of maxillary central incisors.

SECONDARY OUTCOMES:
Lateral negative space | Change from Baseline lateral negative space, at an average 24 months
  The buccal corridor between the posterior teeth and the corner of the mouth in smiling.
Smile arc | Change from Baseline smile arc, at an average 24 months
  Relationship between a hypothetical curve drawn along The edges of the maxillary anterior teeth and the inner contour of the lower lip in the posed smile.
Lip line | Change from Baseline lip line, at an average 24 months
  The height of the upper lip relative to the maxillary central incisors.
Smile width | Change from Baseline smile width, at an average 24 months
  The distance between the most medial points on the lips at the angles of the mouth (Left to right cheilion, CHR to CHL).
Smile height | Change from Baseline smile height, at an average 24 months
  Distance from the most inferior point on the upper lip between the maxillary central inciors to the most superior point on the lower lip on a perpendicular vertical line from the upper point (upper stomion to lower stomion,UST to LST).

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Aboelnaga, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided